CLINICAL TRIAL: NCT05848661
Title: AUDISSEE-Evaluation of a New Digital Therapy of a Cognitive Auditory Training
Brief Title: Evaluation of a Digital Therapy of Auditory Training
Acronym: AUDISSEE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Humans Matter (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-A00248-37
Record Dates: First submitted 2023-03-22; First posted 2023-05-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hearing Loss, Age-Related
Keywords: Hearing aid; presbycusis; auditory training; hearing in noise
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Intervention Model Description: In this study, 240 patients will be randomized in four groups. The first group will be trained with AUDISSEE-verbal, AUDISSE-non-verbal then with the placebo therapy. The second group will be trained with AUDISSEE-non-verbal, AUDISSEE-verbal, then with the placebo therapy. The third group will be trained with the placebo therapy then AUDISSEE-verbal, and AUDISSE-non-verbal. The fourth group will be trained with the placebo therapy then AUDISSEE-non-verbal, and AUDISSE-verbal.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The training will be performed at home. The investigators/evaluators will send a download link of the therapy to the patients without knowing which therapy it corresponds to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AUDISSEE-verbal, AUDISSE-non-verbal, Placebo, Placebo (Experimental): In this arm, the group will perform first the AUDISSEE therapy starting with the verbal sub-training then the non-verbal sub-training. Then it will perform the placebo training for 10 weeks.
  The AUDISSEE therapy takes place over 10 weeks with 3 sessions of 20 minutes per week. It is divided into two parts (5 weeks for each part):
  * verbal training exercises in noise that are specifically aimed at improving patients' intelligibility in noise
  * non-verbal training exercises using environmental sounds and musical sounds, which are specifically aimed at improving non-verbal auditory perception
  Interventions: Device: AUDISSEE; Device: Placebo
- AUDISSE-non-verbal, AUDISSEE-verbal, Placebo, Placebo (Experimental): In this arm, the group will perform first the AUDISSEE therapy starting with the non-verbal sub-training then the verbal sub-training. Then it will perform the placebo training for 10 weeks.
  Interventions: Device: AUDISSEE; Device: Placebo
- Placebo, Placebo, AUDISSEE-verbal, AUDISSE-non-verbal (Placebo Comparator): In this arm, the group will perform first placebo training for 10 weeks. Then, it will perform the AUDISSEE therapy starting with the verbal sub-training then the non-verbal sub-training.
  At each session of the placebo therapy, the patient will listen to an excerpt from an audio-book or podcast of similar length to the duration of the training exercises (20 min).
  This therapy engages the patient in a similar manner than the AUDISSEE therapy in terms of time spent (same session frequency, same session duration), but does not specifically train auditory perception networks.
  Interventions: Device: AUDISSEE; Device: Placebo
- Placebo, Placebo, AUDISSE-non-verbal, AUDISSEE-verbal (Placebo Comparator): In this arm, the group will perform first placebo training for 10 weeks. Then, it will perform the AUDISSEE therapy starting with the non-verbal sub-training then the verbal sub-training.
  Interventions: Device: AUDISSEE; Device: Placebo

INTERVENTIONS:
Device: AUDISSEE — AUDISSEE is a digital therapy designed specifically to improve the hearing in noise of presbycusis patients by offering a complete cognitive auditory training, with verbal and non-verbal stimuli. The therapy takes place over 10 weeks with 3 sessions of 20 minutes per week.
Device: Placebo — The Placebo is a therapy designed within the same frame as the AUDISSEE therapy but with no auditory exercises, instead the patients are listening to audiobook. The therapy takes place over 10 weeks, with 3 sessions of 20 minutes per week.

SUMMARY:
The aim of the study is to evaluate the efficiency of the medical device AUDISSEE in improving the perception in noise ability of presbycusis patients with hearing-aids.

DETAILED DESCRIPTION:
AUDISSEE is a digital therapy designed specifically to improve the hearing in noise of presbycusis patients by offering a complete cognitive auditory training, with verbal and non-verbal (especially musical) stimuli. This therapy is designed improve the comfort of life of people fitted with hearing aids by improving the observance of the wearing of their hearing aids. It is designed for the greatest number of people regardless of age or type of hearing aids and adapts to all levels of hearing loss (mild to severe).

In this study, 240 patients will be randomized in four groups. The first group will be trained with AUDISSEE-verbal, AUDISSE-non-verbal then with the placebo therapy. The second group will be trained with AUDISSEE-non-verbal, AUDISSEE-verbal, then with the placebo therapy. The third group will be trained with the placebo therapy then AUDISSEE-verbal, and AUDISSE-non-verbal. The fourth group will be trained with the placebo therapy then AUDISSEE-non-verbal, and AUDISSE-verbal.

Each training session will last 20 minutes. 3 sessions are planned per week, for 5 weeks for each sub-training. The protocol lasts 20 weeks in total for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* No neurological or psychiatric background
* No major cognitive deficit, able to understand and apply the recommendation
* Motivated to participate
* Have given its written consent
* Affiliated to a social security system
* Diagnostic of presbycusis by a health professional
* Hearing-aids since less than 2 years (no cochlear implants)
* No tinnitus
* With a possible access to a personal computer, tactile tablet or smart-phone to perform the training

Exclusion Criteria:

* Age below 18
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Hearing in noise | 5 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using SpeechNoise and a SNR (Signal-to-Noise Ratio) of 5dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 5 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using CocktailParty noise and a SNR (Signal-to-Noise Ratio) of 10dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 10 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using SpeechNoise and a SNR (Signal-to-Noise Ratio) of 5dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 10 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using CocktailParty noise and a SNR (Signal-to-Noise Ratio) of 10dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 15 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using SpeechNoise and a SNR (Signal-to-Noise Ratio) of 5dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 15 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using CocktailParty noise and a SNR (Signal-to-Noise Ratio) of 10dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 20 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using SpeechNoise and a SNR (Signal-to-Noise Ratio) of 5dB, a percentage of correct repetition of 20 sentences is measured
Hearing in noise | 20 weeks to baseline
  Measure of speech-in-noise comprehension using vocal audiometry (FrBio):
  Using CocktailParty noise and a SNR (Signal-to-Noise Ratio) of 10dB, a percentage of correct repetition of 20 sentences is measured

SECONDARY OUTCOMES:
Quality of life and hearing : personal efficacy | 5 weeks to baseline
  Questionnaire for the feeling of personal efficacy:14 items with a 5-pt likert scale, a mean score is measured (between 1 and 5)
Quality of life and hearing : listening effort | 5 weeks to baseline
  Questionnaire for the listening effort: 10 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing : spatial learning abilities | 5 weeks to baseline
  Questionnaire for the spatial learning abilities (SSQ15): 15 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: personal efficacy | 10 weeks to baseline
  Questionnaire for the feeling of personal efficacy:14 items with a 5-pt likert scale, a mean score is measured (between 1 and 5)
Quality of life and hearing: listening effort | 10 weeks to baseline
  Questionnaire for the listening effort: 10 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: spatial learning abilities | 10 weeks to baseline
  Questionnaire for the spatial learning abilities (SSQ15): 15 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: personal efficacy | 15 weeks to baseline
  Questionnaire for the feeling of personal efficacy:14 items with a 5-pt likert scale, a mean score is measured (between 1 and 5)
Quality of life and hearing: listening effort | 15 weeks to baseline
  Questionnaire for the listening effort: 10 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: spatial learning abilities | 15 weeks to baseline
  Questionnaire for the spatial learning abilities (SSQ15): 15 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: personal efficacy | 20 weeks to baseline
  Questionnaire for the feeling of personal efficacy:14 items with a 5-pt likert scale, a mean score is measured (between 1 and 5)
Quality of life and hearing: listening effort | 20 weeks to baseline
  Questionnaire for the listening effort: 10 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Quality of life and hearing: spatial learning abilities | 20 weeks to baseline
  Questionnaire for the spatial learning abilities (SSQ15): 15 items with a 10-points likert scale, a mean score is measured (between 1 and 10)
Non-verbal auditory testing :pitch change detection task | 5 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Pitch Change Detection task: percentage of correct responses
Non-verbal auditory testing: Direction of pitch change identification task | 5 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Direction of pitch change identification task: percentage of correct responses
Non-verbal auditory testing: Short term memory for pitch task | 5 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Short term memory for pitch task: percentage of correct responses
Non-verbal auditory testing: Emotional prosody recognition task | 5 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Emotional prosody recognition task: perception of correct responses
Non-verbal auditory testing: Auditory Streaming separation task | 5 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Auditory Streaming separation task: mean frequency (in Hz) of perception change between 1 and 2 streams
Non-verbal auditory testing: Pitch Change Detection task | 10 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Pitch Change Detection task: percentage of correct responses
Non-verbal auditory testing: Direction of pitch change identification task | 10 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Direction of pitch change identification task: percentage of correct responses
Non-verbal auditory testing: Short term memory for pitch task | 10 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Short term memory for pitch task: percentage of correct responses
Non-verbal auditory testing: Emotional prosody recognition task | 10 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Emotional prosody recognition task: perception of correct responses
Non-verbal auditory testing: Auditory Streaming separation task | 10 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Auditory Streaming separation task : mean frequency (in Hz) of perception change between 1 and 2 streams
Non-verbal auditory testing: Pitch Change Detection task | 15 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Pitch Change Detection task: percentage of correct responses
Non-verbal auditory testing: Direction of pitch change identification task | 15 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Direction of pitch change identification task: percentage of correct responses
Non-verbal auditory testing: Short term memory for pitch task | 15 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Short term memory for pitch task: percentage of correct responses
Non-verbal auditory testing: Emotional prosody recognition task | 15 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Emotional prosody recognition task: perception of correct responses
Non-verbal auditory testing: Auditory Streaming separation task | 15 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Auditory Streaming separation task : mean frequency (in Hz) of perception change between 1 and 2 streams
Non-verbal auditory testing: Pitch Change Detection task | 20 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Pitch Change Detection task: percentage of correct responses
Non-verbal auditory testing: Direction of pitch change identification task | 20 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Direction of pitch change identification task: percentage of correct responses
Non-verbal auditory testing: Short term memory for pitch task | 20 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Short term memory for pitch task: percentage of correct responses
Non-verbal auditory testing: Emotional prosody recognition task | 20 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Emotional prosody recognition task: perception of correct responses
Non-verbal auditory testing: Auditory Streaming separation task | 20 weeks to baseline
  Battery of listening tests for non-verbal auditory cognition assessment:
  - Auditory Streaming separation task : mean frequency (in Hz) of perception change between 1 and 2 streams

CONTACTS AND LOCATIONS:
Overall Officials: agathe pralus, PhD, Study Chair — Humans Matter

IPD SHARING:
Plan to Share IPD: No